CLINICAL TRIAL: NCT02816437
Title: Fecal Microbiota Transplantation for the Treatment of Multidrug-Resistant Organism Colonization in Solid Organ Transplant Recipients
Brief Title: FMT for MDRO Colonization in Solid Organ Transplant
Acronym: FMT
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: safety
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Lilian Abbo, Associate Profesor of Clinical Medicine, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20160351
Record Dates: First submitted 2016-06-10; First posted 2016-06-28 (Estimated); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Infection Due to Resistant Organism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OpenBiome FMT retention enema (Experimental): OpenBiome Fecal Microbiota Transplantation retention enema, one rectal application.
  Interventions: Biological: OpenBiome Fecal Microbiota Transplantation retention enema

INTERVENTIONS:
Biological: OpenBiome Fecal Microbiota Transplantation retention enema — Keep enema frozen until ready for administration. A single transfer of all 250mL of fecal material using universal precautions to a standard retention enema bag over 1 hour with material retained for at least 1 hour.
  Other Names: Frozen Fecal Enema "OpenBiome"

SUMMARY:
This is a pilot feasibility study to determine whether fecal microbiota transplantation (FMT) can suppress or reverse gastrointestinal carriage of MDROs in hospitalized solid organ transplant recipients with a history of one or more MDRO infections.

DETAILED DESCRIPTION:
This is a pilot feasibility study to determine whether fecal microbiota transplantation (FMT) can suppress or reverse gastrointestinal carriage of MDROs in hospitalized solid organ transplant recipients with a history of one or more MDRO infections.

Study participants who meet inclusion/exclusion criteria and provide written, informed consent will provide a pre-FMT stool sample. Participants will be followed from the time of enrollment up to 3 months post FMT.

Specific organisms of interest that will be tested for by the stool cultures include vancomycin resistant enterococcus, carbapenem resistant Enterobacteriaceae and carbapenem resistant Pseudomonas. Eligible patients who demonstrate colonization with a positive culture for a specific organism of interest will be given FMT.

One FMT dose of a retention rectal enema (OpenBiome) will be administered by a nurse and supervised by our principal investigator and/or sub-investigators trained in performance of FMT.

Stool samples of study participants will be collected and analyzed as follows:

* Pre-FMT: Stool collection & storage in glycerol/flash frozen, to be shipped in dry ice
* 48 hours post FMT: Stool collection using RNA later kit provided by OpenBiome (in hospital)
* Day 7: Stool collection & storage in glycerol/flash frozen, to be shipped in dry ice
* Day 14: Stool collection using RNAlater kit (at home)
* Day 30: Stool collection & storage in glycerol/flash frozen (in hospital or clinic), to be shipped in dry ice
* Day 90: follow-up visit in clinic, final sample collected using RNAlater kit

ELIGIBILITY:
Inclusion Criteria

* Age ≥18 years old
* Solid organ transplant recipients: liver, intestinal, multivisceral transplants, heart, lung, pancreas or kidney transplant recipients
* Transplant recipient at least >30 days post solid organ-transplant
* Transplant recipient must be available locally for follow up to 6-months post FMT transplant
* Inpatient status at time of FMT
* History of at least one or more treated infections in the last 90 days (bacteremia, UTI, pneumonia or abdominal collection with a positive culture with MDRO) due to an MDRO and the MDRO is likely of enteric origin (carbapenem resistant enterobacteriaceae (CRE), vancomycin resistant enterococci (VRE) or carbapenem resistant Pseudomonas (CRP).
* Be without active infection for >15 days: bacteremia, UTI, pneumonia or abdominal collection.
* Be without a positive culture (except for stool) with MDRO (carbapenem resistant enterobacteriaceae (CRE), vancomycin resistant enterococci (VRE) or carbapenem resistant Pseudomonas (CRP)
* Patients are not receiving antimicrobials (therapeutic or suppressive) within 48 hours of FMT
* Solid organ prophylactic antimicrobials as per protocol will be held 24 hours before and 14 days post FMT e.g. trimethoprim/sulfamethoxazole 3x/week or dapsone 100 mg PO daily or weekly for PJP prophylaxis
* Ganciclovir or valgancyclovir for CMV prophylaxis if required as per protocol can be continued.
* Patients have a positive surveillance rectal culture for evidence of colonization.

Exclusion Criteria

* Inability to provide informed consent
* Physician-documented, severe allergy to nuts or other food allergens
* Patients with allergies to ingredients Generally Recognized As Safe " glycerol, sodium chloride
* Study participants hospitalized in the intensive care unit
* CMV IgG, EBV IgG and PCR negative at the time of consent
* Biological MELD score > 28 as defined by transplant surgeon
* Pregnancy or inability/unwillingness to use contraceptives.
* Autoimmune hepatitis
* Patients that received a new solid organ transplant within the last 30 days at the time of enrollment
* Patients on antibiotics treating an active infection or less than 2 weeks at the time of enrollment
* Any circulatory failure on vasopressors
* Respiratory failure (on mechanical ventilation) at the time of enrollment
* Renal failure (GFR <30 or dialysis) at the time of enrollment
* Any active Clostridium difficile infection regardless of severity
* Post-allogeneic hematopoietic stem cell transplant recipients
* ANC <1000/mm3
* HIV+ controlled or not well controlled on antiretroviral therapy
* At increased risk for peritonitis: presence of intra-abdominal devices, peritoneal dialysis.
* Previous FMT
* Patients undergoing treatment for liver or any other organ transplant rejection
* Patients with graft vs. host disease
* Patients with any active infection (bacteremia, pneumonia, urinary tract infection or abscess)
* Life expectancy <1-year post transplant
* Any clinical significant bleeding from a lower GI source (as defined as requiring blood transfusion, endoscopy or surgical or radiologic intervention) in the last 30 days.
* Any condition that the physician investigators deems unsafe, feel the risks of outweigh potential benefit, including other conditions or medications that the investigator determines puts the subject at greater risk from FMT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 10 months
  Overall rates of adverse events

SECONDARY OUTCOMES:
Rate of MDRO decolonization | 10 months
  Number of successful cases of MDRO decolonization
Rate of Recurrent MDRO infections | 10 months
  Number of patients with recurrent MDRO infections

CONTACTS AND LOCATIONS:
Overall Officials: Lilian Abbo, M.D, Principal Investigator — University of Miami

IPD SHARING:
Plan to Share IPD: No